CLINICAL TRIAL: NCT02856750
Title: A Multicenter, Randomized Controlled Trial of the Efficacy of Gabapentin vs. Placebo for Adjuvant Pain Control Following Acute Rib Fractures
Brief Title: Efficacy of Gabapentin vs. Placebo for Adjuvant Pain Control Following Acute Rib Fractures
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-1170
Record Dates: First submitted 2016-07-15; First posted 2016-08-05 (Estimated); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gabapentin (Experimental): gabapentin 300 mg three times daily x 30 d
  Interventions: Drug: Gabapentin
- placebo (No Intervention): no gabapentin administered to this arm.

INTERVENTIONS:
Drug: Gabapentin — Gabapentin 300 mg three times daily x30 days
  Other Names: neurontin
  Arms: gabapentin

SUMMARY:
A Multi-center, Randomized Controlled Trial of the Efficacy of Gabapentin vs. Placebo for Adjutant Pain Control Following Acute Rib Fractures.

DETAILED DESCRIPTION:
Traumatic rib fractures are a tremendous source of pain which can limit respiratory function and overall recovery. Numerous multimodal pain management strategies have been employed with varying success; however, narcotics remain the mainstay of treatment. Beyond the acute side effects of narcotics, including altered mental status, depression of respiratory drive, and constipation, there is a substantial risk of long term dependency. Recently, loco-regional blockade and non-narcotic adjuncts have received increasing support within the literature. Gabapentin has been used extensively as a non-narcotic adjunct to analgesia regimens in the acute and chronic settings, however its ability to better control pain secondary to traumatic rib fractures has never been studied .

The primary aim is to assess the efficacy of gabapentin as an analgesic after rib fractures. Secondary aims are to assess the effect on pulmonary function and other known complications following rib fractures.

The hypothesis is gabapentin will improve pain control as measured by lower pain scores and lower narcotic needs. The investigators plan to test this hypothesis by recruiting trauma patients with rib fractures, and randomly assign them to gabapentin versus a placebo.

ELIGIBILITY:
Inclusion Criteria:

* > 1 rib fractures
* Requiring hospital admission
* Enrolled within 24 hours of injury

Exclusion Criteria:

* Pregnancy
* Intubation
* Age <18, age >65
* Inability to tolerate PO medication
* Patient refusal
* Inability to obtain consent from patient or surrogate
* Renal or Hepatic impairment
* Allergy or Hypersensitivity to gabapentin or any component of the formulation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10-23 (Actual); Study Completion 2018-10-23 (Actual)

PRIMARY OUTCOMES:
Average Daily Pain Score | 30 days
  the pain score uses the visual analog scale and ranges from 0 to 10. This is recorded by nursing at pre-specified intervals depending on level of care.

SECONDARY OUTCOMES:
Narcotic requirements | 30 days
  measurement of daily narcotic use as 24 hour requirements of morphine equivalents, and duration of narcotic needs.
pulmonary function | 30 days
  assessment of the incidence of pneumonia (defined clinically by the treatment team), the incidence of hypoxemia, as well as readmission for pulmonary compromise.

CONTACTS AND LOCATIONS:
Overall Officials: Fredric M Pieracci, MD, PMPH, Principal Investigator — Denver Health
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sirmali M, Turut H, Topcu S, Gulhan E, Yazici U, Kaya S, Tastepe I. A comprehensive analysis of traumatic rib fractures: morbidity, mortality and management. Eur J Cardiothorac Surg. 2003 Jul;24(1):133-8. doi: 10.1016/s1010-7940(03)00256-2. PMID 12853057
- [Background] Chapman BC, Herbert B, Rodil M, Salotto J, Stovall RT, Biffl W, Johnson J, Burlew CC, Barnett C, Fox C, Moore EE, Jurkovich GJ, Pieracci FM. RibScore: A novel radiographic score based on fracture pattern that predicts pneumonia, respiratory failure, and tracheostomy. J Trauma Acute Care Surg. 2016 Jan;80(1):95-101. doi: 10.1097/TA.0000000000000867. PMID 26683395